CLINICAL TRIAL: NCT06671626
Title: Intracranial Recordings to Characterize Action Regulation Mechanisms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cedars-Sinai Medical Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nader Pouratian, Professor & Chair, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2024-0280; 1U01NS132788-01 (NIH)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parkinson's disease patients (Experimental): This group consists of Parkinson's disease patients who are undergoing deep brain stimulation surgery for treatment of their movement disorder. Participants will complete behavioral assessments while receiving subcortical DBS stimulation.
  Interventions: Other: Subcortical Stimulation

INTERVENTIONS:
Other: Subcortical Stimulation — Subcortical simulation of the deep brain stimulation surgery target site will be applied by clinically placed deep brain stimulation electrodes at the previously determined therapeutic setting

SUMMARY:
Humans can rapidly regulate actions according to evolving environmental demands, however, impairments of action regulation have been identified across a number of neurological disorders including Parkinson's Disease (PD). A key component of action regulation is action inhibition that occurs when stopping unwanted or inappropriate actions. There is mounting evidence that action inhibition also plays a critical part in selecting between competing alternative actions and switching to new actions in response to environmental changes. The investigators hypothesize that stop circuitry (involving frontal-subthalamic nucleus (STN) pathways) are involved in inhibiting unselected actions during action selection with competing alternatives (in the absence of overt stopping) and that switching motor plans also engages stopping circuitry (involving prefrontal-STN pathways) for cancelling the ongoing action, before changing to new one. The overall goal is to delineate the neural circuitry underlying a broad array of action regulation functions that involve inhibitory control, how these functions interrelate, and how they are implemented within brain networks. In this research, the investigator will take advantage of the unique opportunity provided by awake deep brain stimulation surgery to learn more about how the brain functions in a diseased state and how deep brain stimulation changes these networks to make movement more normal. The investigator will simultaneously assess cortical and subcortical electrophysiology in relation to clinical symptoms and behavioral measures and in response to deep brain stimulation in patients undergoing Deep Brain Stimulation (DBS) implantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Diagnosis of Parkinson's disease (rigid-akinetic subtype or tremor-dominant) based on presence of at least 2 cardinal PD features (tremor, rigidity, or bradykinesia).
* Clinical indication and decision to proceed with subthalamic nucleus deep brain stimulation implantation.
* L-dopa responsive with clearly defined "on" periods, with at least 30% improvement in UPDRS III scores on vs off medications (with documented ON UPDRS III scores).
* Willingness and ability to cooperate during conscious operative procedure for up to 30 minutes.
* Preoperative MRI without evidence of cortical or subdural adhesions or vascular abnormalities.

Exclusion Criteria:

* Patients with recent use (within one week) of anticoagulant or antiplatelet agent use.
* Neurocognitive testing indicating amnestic cognitive deﬁcits (MOCA < 24).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Cortical ECoG and Subcortical recordings | Intra-operative
  Cortical ECoG and subcortical LFP recordings will occur during DBS implantation surgery during the behavioral assessments
Behavioral assessment | Intra-operative
  Each patient will complete a task that assesses action regulation through a decision making, stopping, and switching task.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes